CLINICAL TRIAL: NCT01837472
Title: Evaluating The Effects of Probiotics on Symptoms of Patients With Irritable Bowel Syndrome
Brief Title: Probiotics in the Treatment of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Gholamrezaei, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 390506
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; Functional gastrointestinal disorders; Gut flora; Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Drug: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Probiotic — Patients in the probiotic group received the probiotic compound Balance® (Protexin Co., Somerset, UK) or similar placebo, twice daily after meal for 14 consecutive days. Balance® capsules contains seven bacteria species including Lactobacillus strains (L. casei, L. rhamnosus, L. acidophilus, and L. bulgaricus), Bifidobacterium strains (B. breve and B. longum), and Streptococcus thermophiles. Total viable count (TVC) is 1 x 108 CFU/per capsule. Other Ingredients are Fructo-oligosaccharide as prebiotic, magnesium stearate, and hydroxypropyl methyl cellulose.
  Arms: Probiotic
Drug: Placebo — Patients in the placebo group received the placebo capsule twice daily after meal for 14 consecutive days.
  Arms: Placebo

SUMMARY:
Evidence have shown benefits of gut flora modulation in treatment of irritable bowel syndrome (IBS), but few reports are available on the effects of multistrain probiotics and there are few reports available in this regard from our society. Thus, we investigated if probiotics are effective in our patients as well. We hypothesize that the multistrain probiotic Balance containing seven bacteria species including Lactobacillus strains, Bifidobacterium strains, and Streptococcus thermophiles reduces the symptoms of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65
* diagnosis of IBS based on the Rome III criteria
* willingness to participate

Exclusion Criteria:

* receiving other probiotics compound during the study
* receiving antibiotics during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Abdominal pain | Up to 6 weeks
  Abdominal pain was assessed by Rome III questionnaire at baseline and then after 6 weeks

SECONDARY OUTCOMES:
Quality of Life | Up to 6 weeks
  Quality of life was assessed by the IBS-QOL questionnaire at baseline and then after 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Somaye Farzamnia, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Department of Gastroenterology, Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Background] Brenner DM, Moeller MJ, Chey WD, Schoenfeld PS. The utility of probiotics in the treatment of irritable bowel syndrome: a systematic review. Am J Gastroenterol. 2009 Apr;104(4):1033-49; quiz 1050. doi: 10.1038/ajg.2009.25. Epub 2009 Mar 10. PMID 19277023